CLINICAL TRIAL: NCT02959645
Title: Assessment of Cortical Network Activities in Cervical Dystonia
Brief Title: Assessment of Brain Activities in Cervical Dystonia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1607M91461
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical Dystonia: patients will have Cervical Dystonia
- Healthy control: Healthy Volunteers

SUMMARY:
To address joint position sense in cervical dystonia patients and how it affects the brain activity.

ELIGIBILITY:
Inclusion Criteria:

* patients having cervical dystonia and aged matched healthy control group

Exclusion Criteria:

* cervical dystonia patients with severe head tremor will be excluded

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cervical dystonia will be recruited from the University of Minnesota's Movement Disorders Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Hand Joint Position Sense | 30 minutes

SECONDARY OUTCOMES:
Brain Signals Recorded via Non-Invasive Surface Electromyography | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Elliott Hall-MSP Lab, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Khosravani S, Buchanan J, Johnson MD, Konczak J. Effect of Neck Botulinum Neurotoxin Injection on Proprioception and Somatosensory-Motor Cortical Processing in Cervical Dystonia. Neurorehabil Neural Repair. 2020 Apr;34(4):309-320. doi: 10.1177/1545968320905799. Epub 2020 Feb 26. PMID 32102606